CLINICAL TRIAL: NCT04670796
Title: A Phase I Study to Compare the Pharmacokinetics, Safety, Tolerability, and Immunogenicity Between HLX02 and Herceptin® (US-licensed and EU-approved Reference Products, Double-blind, Randomized, Parallel-group Part) in Healthy Chinese Male Subjects
Brief Title: A Safety and Pharmacokinetic Study Between HLX02 and Herceptin®(US-licensed and EU-approved) in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX02-HV02
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Healthy
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HLX02 (Experimental): patient receive one dose of HLX02
  Interventions: Drug: HLX02
- EU-sourced Trastuzumab (Herceptin®) (Active Comparator): patient receive one dose of EU-sourced Trastuzumab (Herceptin®)
  Interventions: Drug: EU-sourced Trastuzumab (Herceptin®)
- US-licensed Trastuzumab (Herceptin®) (Active Comparator): patient receive one dose of US-licensed Trastuzumab (Herceptin®)
  Interventions: Drug: US-licensed Trastuzumab (Herceptin®)

INTERVENTIONS:
Drug: HLX02 — subject receive one dose of HLX02
  Arms: HLX02
Drug: EU-sourced Trastuzumab (Herceptin®) — subject receive one dose of EU-sourced Trastuzumab (Herceptin®)
  Arms: EU-sourced Trastuzumab (Herceptin®)
Drug: US-licensed Trastuzumab (Herceptin®) — subject receive one dose of US-licensed Trastuzumab (Herceptin®)
  Arms: US-licensed Trastuzumab (Herceptin®)

SUMMARY:
Randomised, double-blind, parallel group Phase I study to compare PK profiles and to assess the safety and immunogenicity between HLX02 and Herceptin® (U.S. and EU).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed Informed Consent Form
2. Healthy Chinese male (healthy is defined as the fact that no clinically significant abnormalities are identified by medical history, physical examination, vital signs, chest X ray, 12-lead ECG and laboratory tests)
3. Aged ≥ 18 and ≤ 45 years
4. Body mass index (BMI) ≥ 19 and ≤ 28 kg/m2
5. Body weight ≥ 50 and ≤ 80 kg
6. LVEF within normal range as examined through echocardiogram within 14 days prior to randomization (>50%)
7. Immunogenicity (anti-drug [anti-trastuzumab] antibody [ADA]) tested as negative
8. Subject agrees that he and his female spouse/partner use reliable contraceptive methods from the time of administration of study drug until 3 months after the end of study, or subject is infertile

Exclusion Criteria:

1. Any clinically serious disease history or allergic disease, such as hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, mental and nervous diseases and tumor
2. Use of monoclonal antibodies or any biological agent within 6 months prior to the administration of the study drug
3. History of allergic reactions, including allergic reactions caused by any drug or excipient in clinical study
4. Use of any prescription or non-prescription drug or dietary supplement within 5 half lives of such drug or dietary supplement or 2 weeks prior to the administration of the study drug (whichever is longer). The traditional Chinese medicine-based dietary supplement should be discontinued 28 days prior to administration of the study drug
5. Donation of blood within 3 months prior to the administration of the study drug
6. Participation in other clinical studies within 3 months prior to the administration of the study drug
7. Positive test result(s) for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody and treponema pallidum
8. History of drug abuse
9. Inability to follow the protocol requirements, instructions and study limitations as judged by investigators, such as noncooperation, inability to return to the site for follow-up visits or inability to complete the whole clinical study
10. Subject confirmed SARS-CoV-2 infection by appropriate test (including but not limited to nucleic acid test) in screening period

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to infinity (AUCinf) | 57 days

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) | 57 days
time to Cmax (Tmax) | 57 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No